CLINICAL TRIAL: NCT01156077
Title: A Phase 1, Open-Label, Multi-Center, Two-Part, Single-Dose, Parallel Design, Safety, Tolerance, and Pharmacokinetic Study of Orally and Intravenously Administered TR-701 FA in 12 to 17 Year Old Adolescent Patients
Brief Title: Pharmacokinetic (PK) Study of Oral and IV TR-701 FA in Adolescent Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1986-026; TR701-111 (Other: TrisuRX Unique ID)
Record Dates: First submitted 2010-06-11; First posted 2010-07-02 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Bacterial Infection
Keywords: antibiotic; Adolescents receiving antibiotics
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral TR-701 FA (Experimental): Single oral dose of 200 mg TR-701
  Interventions: Drug: TR-701 FA
- IV TR-701 FA (Experimental): Single IV infusion of 200 mg TR-701 FA
  Interventions: Drug: TR-701 FA

INTERVENTIONS:
Drug: TR-701 FA — Oral TR-701 FA 200 mg will be given as a single oral dose
  Arms: oral TR-701 FA
Drug: TR-701 FA — TR-701 FA 200 mg will be given as a single 60 minute IV infusion in 250 cc saline
  Arms: IV TR-701 FA

SUMMARY:
This is an open-label, multi-center, two-part, parallel-design study to assess the PK, safety, and tolerability of TR-701 FA and its active metabolite, TR-700, following a single oral dose (Part A) or IV dose (Part B) of TR-701 FA in 12 to 17 year old adolescent patients.

ELIGIBILITY:
Inclusion Criteria:

* males and females, between 12 and 17 years of age, inclusive;
* receiving prophylaxis for or have a confirmed or suspected infection with Gram positive bacteria and receiving concurrent antibiotic treatment with Gram positive antibacterial activity
* in stable condition
* females must be premenarchal, surgically sterile, abstinent, or practicing an effective method of birth control
* males will either be surgically sterile, abstinent, or practicing an effective method of birth control

Exclusion Criteria:

* relevant history of seizures, clinically significant cardiac arrhythmia, cystic fibrosis, moderate or severe renal impairment, or any physical condition that could interfere with the interpretation of the study results
* any acute or chronic condition that, in the opinion of the Investigator, would limit the patient's ability to complete and/or participate in this clinical study
* physician-diagnosed migraine headaches
* history of infection with hepatitis or other significant hepatic disease
* females who are pregnant or breast feeding

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-06-02 (Actual); Primary Completion 2011-09-24 (Actual); Study Completion 2011-09-24 (Actual)

PRIMARY OUTCOMES:
Adolescent PK | 2 days
  To describe the single-dose pharmacokinetics (PK) of IV and oral TR-701 FA administration in 12 to 17 year old adolescent patients, based on the individual plasma and urine concentration-time data.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Bradley JS, Flanagan SD, Arrieta AC, Jacobs R, Capparelli E, Prokocimer P. Pharmacokinetics, Safety and Tolerability of Single Oral or Intravenous Administration of 200 mg Tedizolid Phosphate in Adolescents. Pediatr Infect Dis J. 2016 Jun;35(6):628-33. doi: 10.1097/INF.0000000000001096. PMID 26910588